CLINICAL TRIAL: NCT00211380
Title: Cognitive Improvement With Aripiprazole (Abilify) in Patients With Schizophrenia, (SFBRI).
Brief Title: Cognitive Improvement With Aripiprazole (Abilify) in Patients With Schizophrenia (SFBRI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was too difficult
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: SAM Technology & The San Francisco Brain Research Institute (Unknown)
Responsible Party: Principal Investigator, James C. Patterson, II, MD. Ph, Professor, Louisiana State University Health Sciences Center Shreveport
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSUHSC #H04-021
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: cognition; schizophrenia; schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: aripiprazole — 10-15 mg daily; if needed dosage may be increased to 30 mg daily after 2 weeks; maintenance 15 mg/day, periodically reassessed.
  Other Names: Abilify

SUMMARY:
This is the sister study to the BMS "Cognitive Improvement with Aripiprazole (Abilify)" study (LSUHSC #H04-022). Evaluation of cognitive ability in patients with schizophrenia or schizoaffective disorder both before and after a switch from risperidone, olanzapine, or risperidone Consta injections to aripiprazole may reveal some of the cognitive changes that correlate with the improved response, better side effect profile, and effects on other components of the negative symptom array. Further, examination of brain functional activity using functional magnetic resonance imaging (fMRI) during an episodic memory task, as well as behavioral performance and associated electroencephalographic (EEG) data of working memory and intermediate term verbal memory collected with the Sustained Attention and Memory Brain Function Test (SAM-BFT), may also provide data showing the neural correlates of these changes in cognition.

DETAILED DESCRIPTION:
* Our long-range goal is to understand how the schizophrenic brain is abnormal, as well as how the function of the brain changes in response to antipsychotic medication, to better understand and effectively treat disorders with these drugs. This information can be used in other disorders as well, as there are many psychiatric disorders that are targeted by the newer atypical antipsychotics.
* The objective of this application, which is the next step in pursuit of our long-range goal, is to compare response on a series of cognitive tests (verbal learning, working memory, and attention) and changes in brain activity in a group of patients with schizophrenia or schizoaffective disorder who are taking risperidone, olanzapine, or risperidone Consta injections and who switch to aripiprazole, and in a group of normal control subjects evaluated twice to control for learning effects.
* The central hypothesis of this application is that patients with schizophrenia or schizoaffective disorder that are taking aripiprazole will have improvements in cognition consistent with the medication's efficacy. We expect that changes in brain activity (from fMRI and EEG) will be correlated with this improvement, as determined by performance on cognitive tests. Further, changes in regional connectivity of affected brain regions will reflect these specific cognitive changes related to aripiprazole.
* The rationale for this proposed study is that, once we have a better understanding of which drugs improve cognition and what brain regions respond differentially to aripiprazole and risperidone, olanzapine, or risperidone Consta, we will have a better understanding of the functional differences tied to the differential actions of the drugs. This is important, because we really don't understand how these medications affect cognition. We are especially well suited to undertake the proposed research as we have access to a large population of patients with schizophrenia or schizoaffective disorder here at our institution.

ELIGIBILITY:
Inclusion Criteria:

Patients (n=10):

* All patients included in the study will have a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of schizophrenia or schizoaffective disorder. Outpatients with schizophrenia (DSM-IV 295.00, 295.10, 295.30, 295.60, 295.90) or schizoaffective disorder (DSM-IV 295.70) will be the primary source of subjects for this project, although inpatients that are being discharged will also be acceptable. All patients will be followed longitudinally.
* Patients who are from 18-65 years of age will be accepted.
* Patients will be screened for medical and psychiatric diagnoses.
* At the time of examination and testing, patients must be stable and taking either olanzapine 10 mg per day for at least two weeks, or at least 2 mg of risperidone per day for at least two weeks, or on risperidone Consta injections (at least 25 mg every two weeks) and not taking an anticholinergic medication for at least one week.
* While recruiting stable patients for this study, this does not necessarily mean free of side effects or free of symptoms of schizophrenia or schizoaffective disorder. Patients that express a desire to switch to aripiprazole may be having side effects, or may be worried that increasing the dose of their current medication may cause side effects.

Controls (n=10):

* The normal control group will provide images of normal response on the behavioral and functional measures, as well as control for the scan-rescan (learning, novelty) effects. They will be matched for age, sex, handedness, and level of education with the patients. They will be screened for medical and psychiatric diagnoses.

Exclusion Criteria:

Patients:

* Any comorbid major psychiatric diagnoses (major depressive disorder, obsessive-compulsive disorder, generalized anxiety disorder, panic disorder, any disorder with psychosis other than those used as inclusion criteria, bipolar disorder).
* Any significant or unstable medical disorder (including unstable or uncontrolled diabetes; long term, severe, or uncontrolled hypertension; or any neurological disorder). Clinical judgment will be used on a case-by-case basis. Special care will be taken in examining patients for metabolic disturbances such as hyperglycemia or hyperlipidemia, due to the increased risk of these problems related to the use of antipsychotics. Patients with clinically unstable and markedly abnormal metabolic profiles will be excluded.
* Active alcohol or substance dependence.
* Significant alcohol or substance abuse in the past six weeks or alcohol or substance dependence in the past year (as defined by DSM-IV).
* Unable to speak, read and understand English, or if the study doctor thinks that the patient cannot follow the study procedures.
* Inability to understand the purpose of the study and give consent.
* Subject is hearing impaired.
* Subject is left-handed.
* Significant abnormalities on physical/neurological examination not consistent with an inclusive diagnosis.
* Current treatment with a classical antipsychotic medication.
* Current treatment with an anticholinergic medication.
* History of adverse response or previous lack of response to aripiprazole.
* Pregnant or lactating women.
* Women of childbearing potential not using medically accepted means of contraception (e.g., intrauterine device [IUD], birth control pills, barrier devices, implanted hormones).
* Handedness will be tracked, and left-handed patients will be excluded due to the small sample size and the variance this will add to cognitive testing.

Controls:

* Current treatment with any psychotropic or anticholinergic medication.
* Any major psychiatric diagnoses (major depressive disorder, obsessive-compulsive disorder, generalized anxiety disorder, panic disorder, any disorder with psychosis, bipolar disorder, attention-deficit/hyperactivity, learning or developmental disorder).
* Any significant medical disorder (including unstable or uncontrolled diabetes; long term, severe, or uncontrolled hypertension; or any neurological disorder). Clinical judgment will be used on a case-by-case basis.
* Any active alcohol or substance dependence in the past six weeks.
* Significant alcohol or substance abuse in the past six weeks, or alcohol or substance dependence in the past year (as defined by DSM-IV).
* Inability to speak, read and understand English, or if the study doctor thinks that the patient cannot follow the study procedures.
* Inability to understand the purpose of the study and give informed consent.
* Significant abnormalities on physical/neurological examination.
* Subject is hearing impaired.
* Subject is left-handed.
* Pregnant or lactating women.
* Women of childbearing potential not using medically accepted means of contraception (e.g., IUD, birth control pills, barrier devices, implanted hormones).
* Dropout criteria: subjects that begin the study and are not able to finish the study will be tracked. Ongoing criteria for termination from the study will include:

  * Adverse events that are intolerable to the patient that prevent continued involvement in the study.
  * New onset medical disorder of such significance as to prohibit further involvement.
  * New onset major psychiatric disorder.
  * Initiation or recurrence of alcohol or substance abuse/dependence.
  * Subject withdraws consent for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
fMRI | at Week 2 and Week 16
SAM-BFT + cognitive tests | at Week 3 and Week 16

CONTACTS AND LOCATIONS:
Overall Officials: James C Patterson, MD, PhD, Principal Investigator — LSU Health Sciences Center-Shreveport/Department of Psychiatry
Locations (1):
- Psychopharmacology Research Clinic, Shreveport, Louisiana, United States